CLINICAL TRIAL: NCT01429233
Title: Real Life Experience of the Use of Isomers as ALENCAL(Levoamlodipine) for Evaluation of Efficacy, Safety and Tolerability in the Management of Cardiovascular Disease in Colombian Patients
Brief Title: Real Life Experience of the Use of Isomers as ALENCAL (Levamlodipine) for Evaluation of Efficacy, Safety and Tolerability in the Management of Cardiovascular Disease in Colombian Patients
Acronym: XPRES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Closter Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: COL-CARDIO-NIS001
Record Dates: First submitted 2011-08-29; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Hypertension
Keywords: Observational; Colombia
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a Phase 4, observational, open study in patients whom their doctor for clinical practice prescribes levamlodipine. No medication was provided by the sponsor. The planned observation time is 8 weeks. The 8 weeks of observation involves an evaluation of baseline followed by information gathered from the assessment visits at week 4 and week 8, or clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose primary physician based on their clinical condition and locally approved use will be eligible to participate in this study, and have been prescribe with Levamlodipine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care adults in Colombia
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Effect of therapy in the management of hypertension and other cardiovascular diseases | 8 weeks
  The change from Baseline in Blood Pressure at 8 weeks will be measure to evaluate th efficacy of the therapy.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 8 weeks
  The number of Participants with Serious and Non- seriuous Adverse Events wil be mesure to evaluate the tolerability and safety profile in 8 weeks follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Country Club Bogota, Bogotá, Colombia